CLINICAL TRIAL: NCT07351682
Title: Antibacterial Efficacy of Calcium Hydroxide Used Alone or in Combination With Iodoform (Metapex) and Steroid (Betamethasone) in Patients With Apical Periodontitis
Brief Title: Antibacterial Activity of Calcium Hydroxide and Betamethasone in Apical Periodontitis
Status: Not yet recruiting | Type: Observational
Sponsor: Duygu Degirmencioglu (Other)
Responsible Party: Sponsor-Investigator, Duygu Degirmencioglu, Duygu Degirmencioglu, Medipol University
Organization: Medipol University (Other)
Other Study IDs: MedipolU-629
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Apical Periodontitis
Keywords: Betamethasone; Calcium Hydroxide; Enterococcus faecalis; Droplet Digital PCR; Retreatment
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Intracanal samples will be collected from root canals using sterile paper points during different stages of endodontic retreatment. The samples will contain microbial material from the root canal system and will be used for DNA extraction and molecular analysis. Specimens will be stored under appropriate laboratory conditions until droplet digital PCR (ddPCR) analysis is performed to quantify total bacterial load and Enterococcus faecalis levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Calcium Hydroxide: This cohort includes patients with apical periodontitis undergoing endodontic retreatment who receive calcium hydroxide as an intracanal medicament as part of routine clinical care. The selection of the intracanal medicament is based on standard clinical decision-making and is not assigned by the study protocol.
- Calcium Hydroxide + Iodoform (Metapex): This cohort includes patients with apical periodontitis undergoing endodontic retreatment who receive a combination of calcium hydroxide and iodoform (Metapex) as an intracanal medicament as part of routine clinical care. The intracanal medicament is selected according to standard clinical practice and is not assigned by the study protocol.
- Calcium Hydroxide + Betamethasone: This cohort includes patients with apical periodontitis undergoing endodontic retreatment who receive a combination of calcium hydroxide and betamethasone as an intracanal medicament as part of routine clinical care. The choice of intracanal medicament is determined by routine clinical decision-making and is not assigned by the study protocol.

SUMMARY:
Apical periodontitis is a chronic inflammatory disease caused by bacterial infection of the root canal system. Although mechanical cleaning and shaping reduce most microorganisms, bacteria may persist in areas that are difficult to reach, making the use of intracanal medicaments between treatment sessions clinically important.

Calcium hydroxide is one of the most commonly used intracanal medicaments because of its antibacterial properties. However, some resistant microorganisms, such as Enterococcus faecalis, may survive when calcium hydroxide is used alone. Therefore, combining calcium hydroxide with other agents, such as iodoform or corticosteroids, may improve its antibacterial effectiveness.

The purpose of this study is to compare the antibacterial activity of calcium hydroxide used alone or in combination with iodoform (Metapex) or betamethasone in patients with apical periodontitis. Bacterial load in root canals will be evaluated using droplet digital PCR (ddPCR), a highly sensitive molecular method that allows absolute quantification of bacteria. The results of this study are expected to provide evidence to support optimal intracanal medicament selection in endodontic retreatment cases.

DETAILED DESCRIPTION:
Apical periodontitis is a chronic inflammatory condition of periapical tissues that develops as a result of persistent bacterial infection within the root canal system. While chemomechanical preparation significantly reduces the microbial load, bacteria may remain in anatomical complexities such as dentinal tubules, isthmuses, and apical ramifications. For this reason, intracanal medicaments are widely used between treatment sessions to enhance disinfection and improve treatment outcomes.

Calcium hydroxide is the most frequently used intracanal medicament due to its high pH and antibacterial properties. Nevertheless, certain microorganisms, particularly Enterococcus faecalis, have been shown to survive in alkaline environments, limiting the effectiveness of calcium hydroxide when used alone. To overcome this limitation, calcium hydroxide has been combined with various agents, including iodoform and corticosteroids, with the aim of enhancing antibacterial activity and reducing periapical inflammation.

Droplet digital PCR (ddPCR) is a novel molecular technique that enables absolute quantification of bacterial DNA without the need for standard curves and is less affected by PCR inhibitors compared to conventional quantitative PCR methods. Despite its advantages, the use of ddPCR in clinical endodontic research remains limited, particularly in in vivo studies evaluating intracanal medicaments.

This prospective, single-center clinical study aims to compare the antibacterial efficacy of three intracanal medicament protocols in patients with apical periodontitis undergoing endodontic retreatment: (1) calcium hydroxide alone, (2) calcium hydroxide combined with iodoform (Metapex), and (3) calcium hydroxide combined with betamethasone. Root canal samples will be collected at different treatment stages, and total bacterial load as well as Enterococcus faecalis levels will be quantified using ddPCR.

The findings of this study are expected to provide high-quality clinical evidence regarding the antibacterial effectiveness of commonly used intracanal medicaments and their combinations. The results may contribute to evidence-based decision-making in the selection of intracanal medicaments for the management of apical periodontitis, particularly in retreatment cases.

ELIGIBILITY:
Inclusion Criteria:

* - Adults aged 18 to 65 years.
* Patients diagnosed with apical periodontitis requiring endodontic retreatment.
* Presence of a single tooth with radiographic evidence of apical periodontitis.
* Ability to provide written informed consent.

Exclusion Criteria:

* Use of systemic antibiotics within the previous 3 months.
* Presence of systemic diseases that may affect healing or immune response.
* Pregnancy or lactation.
* Known allergy or hypersensitivity to any of the intracanal medicaments used.
* Teeth with acute abscess, severe periodontal disease, or root fractures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with apical periodontitis who require endodontic retreatment and are treated at a single academic dental center.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Total Bacterial Load in Root Canal Samples | From baseline to 7 days after intracanal medicament application
  The primary outcome is the change in total bacterial load in root canal samples collected during endodontic retreatment. Bacterial load will be quantified using droplet digital PCR (ddPCR) by measuring absolute bacterial DNA copy numbers at different treatment stages.

SECONDARY OUTCOMES:
Change in Enterococcus faecalis Levels | From baseline to 7 days after intracanal medicament application
  This secondary outcome assesses the change in Enterococcus faecalis levels in root canal samples collected during endodontic retreatment. Enterococcus faecalis DNA will be quantified using droplet digital PCR (ddPCR) by measuring absolute DNA copy numbers before and after intracanal medicament application.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Faculty of Dentistry, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No